CLINICAL TRIAL: NCT05299671
Title: Pilot Study to Assess Feasibility of a Pharmacist-Led Video Consultation to Reduce Drug Interactions Among Patients Initiating Oral Anti-Cancer Drugs
Brief Title: Video Consultation to Reduce Drug Interactions Among Patients Initiating Oral Anti-Cancer Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAT3167
Record Dates: First submitted 2022-01-25; First posted 2022-03-29 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video consultation group (Experimental): Patients starting a new oral anti-cancer drug (OACD) will receive help to identify and manage potential drug-drug interactions alongside patient's oncologist through a one-time video consultation.
  Interventions: Behavioral: Video consultation

INTERVENTIONS:
Behavioral: Video consultation — During the video visit, a pharmacist will speak with the patient about potential drug-drug interactions between the patient's cancer treatment and the other medications on the list, make recommendations about medication management (which will also be directly communicated to the oncologist), provide education about the patient's new OACD, and answer any questions. The virtual consultation will last about 30 minutes via an electronic device.

SUMMARY:
This is a non-randomized prospective pilot intervention study to assess the feasibility of a onetime pharmacist-led video consultation for medication review and patient education among patients initiating an oral anti-cancer drug. In addition, investigator will evaluate reductions in polypharmacy, potential DDIs, and patient self-efficacy by comparing these variables for each patient before and after the video consultation.

DETAILED DESCRIPTION:
In this study, the investigator will be evaluating a 30-minute pharmacist-led video consultation to provide education about patients new oral anti-cancer drug (OACD) and help identify and manage potential drug-drug interactions alongside your oncologist. While OACDs offer both clinical benefits and added convenience when compared to traditional intravenous chemotherapy, they also present a number of potential challenges. One critical challenge involves the increased risk of taking multiple oral medications daily. Patients taking multiple medications can result in harmful effects due to unexpected drug interactions, as well as patient confusion regarding when to take specific medications. Given the relatively recent rise in available OACDs, little is known about the extent of this issue

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 years
* Patients must have access to a smartphone, tablet, or computer to facilitate a video visit, or be willing to come into the hospital to borrow a tablet for the visit
* Patients must have received a prescription for a new oral anti-cancer drug within 4 weeks of enrollment, not administered as part of a clinical trial
* Patients must take at least three prescribed, standing oral medications in addition to their newly prescribed anti-cancer drug

Exclusion Criteria:

* Patients who do not speak English or Spanish
* Patients without cognitive capacity to give informed consent for participation
* Patients uncomfortable with using video-based technology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects enrolled that complete the 30 minutes consultation and assessments | 30 minutes
  To determine feasibility of a one-time pharmacist-led video consultation among advanced cancer patients initiating oral anti-cancer drugs. Feasibility will be defined as significant evidence that 50% of enrolled patients will complete all components of the study.
Rate of absorption interaction | Baseline
  Based on the pre-consultation medication reconciliation, we will assess the characteristics (absorption interaction) of medication list inaccuracies identified by medication reconciliation among study participants.
Average of QTc prolongation | Baseline
  Based on the pre-consultation medication reconciliation, we will assess the characteristics ( QTc prolongation) of medication list inaccuracies identified by medication reconciliation among study participants.

SECONDARY OUTCOMES:
Mean of medication list inaccuracies among study participants prior to the consultation | Baseline
  Based on the pre-consultation medication reconciliation, we will assess the mean number of medication list inaccuracies identified by medication reconciliation among study participants.
Change in assess factors associated with OACD-related potential drug-drug interactions and medication inaccuracies | Within 30 days of the consultation
  We will assess patient-level factors associated with OACD-related potential DDIs and medication inaccuracies, such as age, race/ethnicity, socioeconomic status, cancer diagnosis, number of medications, and number of comorbidities.
Number of medication changes recommended | Within 30 days of the consultation
  The number of medication changes recommended to address polypharmacy and/or DDIs
Change in the proportion of patients with a mitigated DDI | Within 30 days of the consultation
  The proportion of patients with a mitigated DDI, defined as a change in one involved medication within 30 days of the consultation
Change in proportion of patients with a reduction in total number of medications and/or supplements | Within 30 days of the consultation
  The proportion of patients with a reduction in total number of medications and/or supplements within 30 days of the consultation
Change in Medication Regimen Complexity Index (MRCI) before and after the consultation | within 30 days of the consultation
  The change in medication list complexity using the Medication Regimen Complexity Index (MRCI) within 30 days of the consultation
Mean Score to Medication Self-Efficacy Scale (MASES) to assess patient confidence and competence regarding OACD administration before and after the consultation | Within 30 days of the consultation
  The change in patient confidence and competence regarding OACD administration using a modified version of the Medication Adherence Self-Efficacy Scale (MASES-R) before and after the consultation
Change in mean score on the Satisfaction with Information about Medications Scale (SIMS) before and after the consultation | Within 30 days of the consultation
  Patient reported outcomes as measured by the Satisfaction with Information about Medications Scale (SIMS)
Change in mean score on the Acceptability of Intervention Measure (AIM) before and after the consultation | Within 30 days of the consultation
  Patient reported outcomes as measured by the Acceptability of Intervention Measure (AIM)
Change in mean score on the Intervention Appropriateness Measure (IAM) before and after the consultation | Within 30 days of the consultation
  Patient reported outcomes as measured by the Intervention Appropriateness Measure (IAM)
Change in mean score on the Feasibility of Intervention Measure (FIM) before and after the consultation | Within 30 days of the consultation
  Patient reported outcomes as measured by the Feasibility of Intervention Measure (FIM)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States